# **Official Title:** Improving Symptom Management for Adolescents and Young Adults With Advanced Cancer: Development and Pilot Testing of a Novel Intervention

**NCT:** NCT05593016

**IRB Document Date:** 5/16/2024

Please read the following information carefully. Please do not skip any sections. If you agree to participate in the research study, you will be asked to indicate this at the end of the document. In order to participate, you as the study participant must give consent.

If you have any questions, please call [Study Staff Name] at [Study Staff Phone Number].

### Consent to Participate in a Research Study

AYA Symptom Management

#### CONCISE SUMMARY

The purpose of this research study is to gain a better understanding of the experiences of adolescents and young adults (aged 15-29) who have been diagnosed with cancer.

You will be asked to complete a baseline assessment and two follow-up assessments over approximately 2.5 months. Each of these assessments will include the completion of surveys. At the end of the baseline assessment, you will be randomized (like the flip of a coin) to either a Symptom Management Program or to the control group that will receive educational materials. The Symptom Management Program includes four individual sessions held over Zoom over a 4-6 week period.

There are minimal risks associated with this study. The greatest risks of this study include loss of confidentiality. Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of the questions. There is also the potential risk of loss of confidentiality, though every effort will be made to keep your information confidential.

If you are interested in learning more about this study, please proceed to the next page.

| I have | e read | the concise | summary | and I wi | ish to co | ontinue | reading the | consent form | n. |
|---|---|---|---|---|---|---|---|---|---|
| I have | e read | the concise | summary | and I Do | O NOT | wish to | participate | in the study | |

If the person chooses not to participate, provide a message that says: "Thank you for your time. You have chosen not to participate in this research study. If you have any questions, please contact the research study team by phone at [study staff phone number] or email [study staff email address]."

# Consent to Participate in a Research Study

**AYA Symptom Management** 

You are being asked to take part in this research study because you have been diagnosed with cancer. Research studies are voluntary and include only people who choose to take part. Please read this consent form carefully and take your time making your decision. As the study doctor or study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. We encourage you to talk with your family and friends before you decide to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below.

DUHS IRB IRB NUMBER: Pro00110574

Please tell the study doctor or study staff if you are taking part in another research study.

A grant from the National Institutes of Health (NIH) will sponsor this study. Portions of Caroline Dorfman, PhD and her research team's salaries will be paid by this grant.

# WHO WILL BE MY DOCTOR ON THIS STUDY?

If you decide to participate, you will not have a different medical doctor. Your regular doctor will continue to be your doctor throughout the time you are in the study. Dr. Caroline Dorfman in the Department of Psychiatry and Behavioral Sciences is conducting this study, and she will be in contact with your regular health care provider throughout the time that he/she is in the study and afterwards, if needed.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this study is to aid in the development of an intervention aimed to improve symptom management for adolescents and young adults with cancer and to examine the impact of the intervention.

# HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Approximately 40 people will take part at in this study at Duke.

#### WHAT IS INVOLVED IN THE STUDY?

If you agree to be in this study, you will be asked to sign and date this consent form. Your medical record will be reviewed to obtain information about your cancer, treatments related to your cancer, and other health conditions. No tests or procedures are required to meet eligibility.

In this study, you will be randomly assigned (like the flip of a coin) to receive a Symptom Management Program or to receive educational materials tailored to the experiences of individuals with cancer. If you are randomized to receive the Symptom Management Program, you will participate in four, 60-minute sessions held over Zoom over a 4-6 week period. You can access Zoom on a study iPad or on your own personal device.

All participants will complete an initial assessment and follow-up assessments approximately 6 and 10 weeks later. You will be given the option to complete assessments on a study iPad or on your own personal devices. During each assessment, you will answer questions about topics including your sociodemographic characteristics, medical history, pain, fatigue, psychological distress, symptom severity and interference, self-efficacy for managing symptoms, and values. Assessments will take approximately 25 minutes to complete

We will send you automated text messages throughout this study. To do this we use a web-based system, called Twilio, which uses your phone number to send you messages. We plan to use this feature to send you text message reminders throughout the study to complete study assessments and study sessions, if relevant. If you agree to receive text message reminders, we will contact you this way during the study. If you change your mind about the messages or if your contact phone number changes, please contact the study team. These messages are one-way only, so you cannot reply. If you have questions or concerns about information in a message, contact your study team.

DUHS IRB

IRB NUMBER: Pro00110574

The Symptom Management Program Zoom sessions will be audio/video recorded. The audio/video recording will be reviewed by members of the study team. Participation in this study is voluntary. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled.

#### HOW LONG WILL I BE IN THIS STUDY?

You will be in the study for approximately 10-12 weeks.

You can choose to stop participating at any time without penalty or loss of any benefits to which you are entitled. However, if you decide to stop participating in the study, we encourage you to talk to your doctor first.

#### WHAT ARE THE RISKS OF THE STUDY?

There are minimal risks associated with this study. Some of the questions we will ask you as a part of the study may make you feel uncomfortable. You may refuse to answer any of the questions. If you are randomized to receive the Symptom Management Program, it is possible that some of the topics discussed may make you feel uncomfortable. Discussing your health or stressors associated with your health may be upsetting. You may choose to not discuss concerns that you find upsetting. Also, you may stop your participation in this study at any time. There is also the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential, however, this cannot be guaranteed.

Many companies and applications on your smartphone commonly use text platforms and cloud-based companies to send and receive information. We use Twilio to send you text messages. Twilio does encrypt your information on their servers, but no system is completely safe. If they decide to share these data, it may no longer be covered under the privacy protections. Information that identifies you, such as your phone number, may be sent to and permanently kept by Twilio and their business associates. Information disclosed to these companies or their business partners may no longer be covered under the privacy protections. Because text messaging does not provide a completely secure and confidential means of communication, if you wish to keep your communication completely private please let us know and we will communicate with you only through regular channels like the telephone and email.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

Participation in this study may provide you with an opportunity to learn skills that can help you better manage symptoms or improve your overall health. We expect that the information learned from this study will benefit other adolescent and young adult cancer patients in the future.

#### WILL MY INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information in order to conduct the research. Your personal information may also be given out if required by law.

DUHS IRB

IRB NUMBER: Pro00110574

Study records that identify you will be kept confidential as required by law. Federal Privacy Regulations provide safeguards for privacy, security, and authorized access. Except when required by law or for your care, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier in study records disclosed outside of Duke University Health System (DUHS). For records disclosed outside of DUHS, you will be assigned a unique code number. The key to the code will be kept securely at DUHS.

If you are randomized to the intervention arm, you will be identified in the audio/video recordings by your study ID number. Any link to your name will be kept in a password protected computer database kept separate from other study data. All recordings will be stored in a password protected computer file on an encrypted laptop and a DUHS secure server. Audio recordings will be available only to authorized study personnel as necessary for the purposes of this study and will be identified by your study ID number. After the study has been completed, all audio recordings will be destroyed.

The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your privacy. With this Certificate, the investigators may not disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use. Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:

- 1) there is a law that requires disclosure (such as to report child abuse or communicable diseases but not for legal proceedings);
- 2) you have consented to the disclosure, including for your medical treatment; or
- 3) the research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project or for information that is required by the Food and Drug Administration (FDA).

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy. Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your name or other personal information will not be revealed.

The study results will be retained in your research record for at least six years after the study is completed. At that time, either the research information not already in your medical record will be destroyed or information identifying you will be removed from such study results at DUHS. Any research information in your medical record will be kept indefinitely.

DUHS IRB IRB NUMBER: Pro00110574

Some people or groups who receive your health information might not have to follow the same privacy rules. Once your information is shared outside of DUHS, we cannot guarantee that it will remain private. If you decide to share your private information with anyone not involved in the study, the federal law designed to protect your health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

#### WHAT ARE THE COSTS TO YOU?

There will not be any cost to you as a result of participating in this study.

#### WHAT ABOUT COMPENSATION?

You will be reimbursed up to \$60 for your expenses related to participation (e.g., time). This reimbursement will consist of \$20 for completing each of the study assessments. If you choose to withdraw from the study, you will only receive compensation for the parts of the study that you completed.

#### WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that you are injured as a result of your participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your Duke physicians to provide monetary compensation or free medical care to you in the event of a study-related injury.

For questions about the study or research-related injury, contact Dr. Caroline Dorfman, PhD at during regular business hours, after hours, and on weekends and holidays.

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You may choose not to be in the study, or, if you agree to be in the study, you may withdraw from the study at any time. If you withdraw from the study, no new data about you will be collected for study purposes other than data needed to keep track of your withdrawal. All data that have already been collected for study purposes will be sent to the study sponsor.

Your decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you are entitled, and will not affect your access to health care at Duke. If you do decide to withdraw, we ask that you contact Dr. Caroline Dorfman in writing and let her know that you are withdrawing from the study. Her email address is caroline.dorfman@duke.edu.

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study.

Your doctor may decide to take you off this study if your condition gets worse, if you have serious side effects, or if your study doctor determines that it is no longer in your best interest to

DUHS IRB

IRB NUMBER: Pro00110574

continue. The sponsor or regulatory agencies may stop this study at anytime without your consent. If this occurs, you will be notified and the study team will discuss other options with you.

A description of this study will be available on <a href="https://www.clinicaltrials.gov/">https://www.clinicaltrials.gov/</a> as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, contact Dr. Caroline Dorfman at during regular business hours, after hours, and on weekends and holidays.

For questions about your rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.

#### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form."

DUHS IRB IRB NUMBER: Pro00110574